CLINICAL TRIAL: NCT04072562
Title: An Open-label, Single-centre, Randomised, 3-period, 3-treatment, Single-dose, Crossover Study to Assess the Relative Bioavailability of AZD7594 Inhaled Via a Nebulizer and Via a Dry Powder Inhaler in Healthy Subjects
Brief Title: A Study to Evaluate the Amount of Drug That Becomes Available to the Blood Circulation When Inhaled by a Nebulizer and Dry Powder Inhaler in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3742C00001
Record Dates: First submitted 2019-07-19; First posted 2019-08-28 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Asthma
Keywords: Bioavailability; Pharmacokinetics; Safety; Selective glucocorticoid receptor modulator
MeSH Terms: conditions — Asthma | interventions — velsecorat

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AZD7594 0.7 mg (Experimental): The study subjects will receive AZD7594 via nebulizer, during 8 minutes: 0.7 mg, delivered dose 1 inhalation
  Interventions: Drug: AZD7594
- AZD7594 1.6 mg (Experimental): The study subjects will receive AZD7594 via nebulizer, during 8 minutes: 1.6 mg, delivered dose 1 inhalation
  Interventions: Drug: AZD7594
- AZD7594 720 μg (Active Comparator): The study subjects will receive AZD7594 via DPI: 0.72 mg, delivered dose (792 µg nominal dose) 1 inhalation
  Interventions: Drug: AZD7594

INTERVENTIONS:
Drug: AZD7594 — Treatment A: The study drug is a nebulizer suspension with strength 2.8 mg/mL using 2 mL in the device. The study drug is administered via oral inhalation.
  Treatment B: The study drug is a nebulizer suspension with strength 6.3 mg/mL using 2 mL in the device. The study drug was administered via oral inhalation.
  Treatment C: The study drug is an inhalation powder. The study drug was administered via oral inhalation.

SUMMARY:
The purpose of this study is to assess the relative bioavailability of the AZD7594 nebulized formulations (test) and the dry powder formulation (reference).

The study results will provide information on the pharmacokinetic (PK) profile following use of the 2 devices to be used in further clinical development.

DETAILED DESCRIPTION:
This study will be an open-label, randomised, 3 period, 3-treatment, crossover study in healthy subjects (males and females), performed at a single clinical unit.

The study will comprise:

* A screening period of maximum 28 days;
* Three treatment periods during which subjects will be resident from the morning (fasting conditions) of the day before dosing with AZD7594 (Day -1) until at least 48 hours after dosing; discharged on the morning of Day 3;
* Two ambulatory visits (Day 4 and Day 5) within each treatment period; and
* A final visit 10 to 14 days after the last administration of AZD7594.
* There will be a minimum washout period of 10 days between each dose administration.

A total of 24 subjects will be randomised to receive single doses of AZD7594 on 3 occasions, under fasted conditions (overnight fast of at least 10 hours):

* Treatment A: 0.7 mg (delivered dose) AZD7594 via nebulizer, test
* Treatment B: 1.6 mg (delivered dose) AZD7594 via nebulizer, test
* Treatment C: 720 μg (delivered dose) AZD7594 via dry powder inhaler (DPI), reference

Each subject will be involved in the study for approximately 10 to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female subjects aged 18 - 55 years (inclusive) at Screening with suitable veins for cannulation or repeated venepuncture.
3. Females must have a negative pregnancy test at screening and on admission to the unit for each treatment period, and must not be lactating. Women of child-bearing potential (WOCBP) must be stable on their chosen method of highly effective birth control for a minimum of 3 months prior to Visit 1, and willing to use that for the entire duration of the study (from the time they sign the informed consent), and for 14 days after the last dose of IMP. They must agree not to become pregnant or donate ova throughout the study and for 14 days after the last dose of IMP. Male subjects must be surgically sterile or be willing to use a condom during the study.
4. Have a body mass index (BMI) between 18 and 29.9 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive).
5. Subject is able to understand and communicate in German.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. History of Gilbert's syndrome, history of cholecystectomy or gall stone.
4. History of tuberculosis, any other significant lung diseases like surgeries, asthma, chronic obstructive pulmonary disease.
5. Upper respiratory tract infections (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within 3 months prior to Screening.
6. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
7. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, at screening and first admission to the study unit (first treatment period) as judged by the PI.
8. Any clinically significant abnormal findings in vital signs at screening and first admission to the study unit (first treatment period), as judged by the PI, and defined as:

   * Systolic BP <90 mmHg or ≥140 mmHg and diastolic BP <50 mmHg or ≥90 mmHg
   * Heart rate <50 bpm or >90 bpm
9. Any clinically significant abnormalities on 12-lead ECG at screening and first admission to the study unit (first treatment period), as judged by the PI, and defined as:

   * Sick sinus syndrome
   * Arrhythmia
   * Prolonged QT interval corrected using Fridericia's formula > 450 ms
10. Any positive result at screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) results.
11. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomised in this study or other clinical studies, are not excluded.
12. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
13. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity to AZD7594 or formulation excipients, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7594.

    Note: subjects with hay fever are allowed to participate, unless hay fever is active
14. Current smokers or those who have smoked or used nicotine products (including e-cigarettes; >10 pack-year) within the 6 months prior to screening.
15. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the PI or positive screen for drugs of abuse, cotinine, and/or alcohol at screening or on each admission to the clinical unit.
16. Use of drugs with enzyme-inducing properties within 3 weeks prior to the first administration of IMP or herbal preparations/medications including, but not limited to, St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng. Subjects should stop using these herbal medications 14 days prior to the first administration of IMP.
17. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life.

    Note: Hormonal replacement therapy (HRT) and systemic contraceptives are allowed for females.
18. Subjects not able to perform a technically acceptable spirometry and/or not able to use the DPI correctly or not able to tolerate the pre-defined inhalation/nebulization.
19. Subjects with a pregnant partner.
20. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
21. Subjects who have previously received AZD7594.
22. Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL
Area under plasma concentration-time curve from zero to infinity (AUC) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC0-t) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL
Individual ratios of test versus reference for AUC | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL
Individual ratios of test versus reference for AUC0-t | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL
Individual ratios of test versus reference for Cmax | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To estimate the relative bioavailability of AZD7594 following inhalation via nebulizer Omron NE C900-E (2 dose levels) and via DPI SD3FL

SECONDARY OUTCOMES:
Time to reach maximum observed plasma concentration (tmax) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Terminal elimination rate constant (λz) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Half-life associated with terminal slope (λz) of a semilogarithmic concentration-time curve (t1/2λz) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Mean residence time of the unchanged drug in the systemic circulation from zero to infinity (MRT) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | At pre-dose, at 15, 30, and 45 minutes, and at 1, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post dose (Days 1, 2, 3, 4 and 5)
  To evaluate the PK profiles of AZD7594 when administered as the two formulations
Number of participants with adverse events | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in systolic BP | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in diastolic BP | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in pulse rate | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in body temperature | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in ECG | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in physical examination | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers. The complete physical examinations will include an assessment of the general appearance, respiratory, cardiovascular, abdomen, skin, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems.
Number of participants with abnormal findings in spirometry | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers. All spirometry measurements will be performed using the Jaeger Masterscope for which calibration will be performed daily using a 3 L calibration syringe. Spirometry measurements with the Jaeger Masterscope will be performed according to European Respiratory Society/American Thoracic Society guidelines. Global Lung Function Initiative 2012 reference values will be used.
Number of participants with abnormal findings in haemoglobin | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in haematocrit | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in white blood cell count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in red blood cell count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in mean corpuscular volume (MCV) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in mean corpuscular haemoglobin (MCH) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in mean corpuscular hemoglobin concentration (MCHC) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in neutrophils absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in lymphocytes absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in monocytes absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in eosinophils absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in basophils absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in platelets | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in reticulocytes absolute count | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers
Number of participants with abnormal findings in sodium | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in potassium | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in urea | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in creatinine | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in albumin | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in calcium | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in phosphate | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in glucose (fasting) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in C-reactive protein | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in T4 hormone | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in thyroid-stimulating hormone | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in liver enzymes | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers. The laboratory variables to be measured are: Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma glutamyl transpeptidase (GGT)
Number of participants with abnormal findings in total bilirubin (TBL) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in unconjugated bilirubin | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in follicle stimulating hormone (FSH) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in lutenizing hormone (LH) | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers.
Number of participants with abnormal findings in coagulation | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers. The laboratory variables to be measured are: international normalized ratio and activated partial thrombin time
Number of participants with abnormal findings in urinalysis | From Screening (Day -28) up to the Follow-up visit (10 to 14 days after last dose)
  To further assess the safety of single doses of AZD7594 in healthy volunteers. The laboratory variables to be measured are: protein, glucose, and blood.

OTHER OUTCOMES:
AZD7594 concentrations in dried blood PK sample | Days 1, 2 and 3 (2, 6, 12, 24 and 48 h post dose)
  To assess AZD7594 concentrations in dried blood PK samples (collected via both venepuncture and finger prick) and compare with wet blood and plasma PK samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, Principal Investigator — Parexel
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No